CLINICAL TRIAL: NCT01460121
Title: A Randomized, Double Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of SpotOn Specs™ for the Treatment of Chronic Dizziness
Brief Title: Study to Assess the Efficacy and Safety of SpotOn Specs™ for the Treatment of Chronic Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Collaborators: SpotOn Therapeutics Ltd. (Industry)
Responsible Party: Principal Investigator, carlos gordon, Professor, Department of Neurology, Meir Medical Center, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SpotOn Specs 002
Record Dates: First submitted 2011-10-25; First posted 2011-10-26 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Chronic Dizziness
Keywords: Phobic Postural Vertigo; Visual Vertigo; Chronic Subjective Dizziness; Motion and Space Discomfort; SpotOn

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SpotOn's corrective elements (Experimental)
  Interventions: Device: SpotOn's corrective elements for dizziness
- Placebo corrective elements (Placebo Comparator)
  Interventions: Device: SpotOn's corrective elements for dizziness; Device: Placebo

INTERVENTIONS:
Device: SpotOn's corrective elements for dizziness — Eyeglasses with dizziness correction elements (real SpotOn eyeglasses) or eyeglasses with placebo (sham eyeglasses) elements will be worn during the whole four weeks study period.
Device: Placebo
  Arms: Placebo corrective elements

SUMMARY:
The diagnosis and management of acute vertigo and dizziness is most of the time an easy task for the general practitioner. However, following an acute vestibular disorder and very often with no any overt cause, a considerable number of patients complain on chronic dizziness and subjective disturbance of balance despite normal clinical and laboratory tests. Patients describe that perceptual visual stimulus provoke or aggravate their symptoms that are frequently accompanied by anxiety. These cases have been described in the medical literature as Phobic Postural Vertigo, Visual Vertigo, Chronic Subjective Dizziness and Motion and Space Discomfort (2,3,4,5). Treatment of these conditions includes physical therapy (similar to vestibular rehabilitation exercises) and anti-anxiety or anti-depressant agents such as benzodiazepines and SSRI, however, the effectiveness of these approaches is debatable.

Because visual stimuli play a crucial role in space orientation and motion perception, it is reasonable to hypothesize that certain visual stabilizing signals applied on the peripheral visual field (that is involved mainly in the perception of motion) could be of help in patients suffering from dizziness. This is the rationale of a new technology (SMB- Senso Mental Balance Technology) developed to alleviate the feelings of dizziness.

Trial is conducted in Meir Medical Center, Israel. Recruitment only in Israel!

ELIGIBILITY:
Inclusion Criteria:

* Age: 18≤ years ≤85
* Clinical diagnosis of chronic dizziness primary or secondary to vestibular disorder.
* Stable symptoms for more than one month and less than a year.
* Ability to perform all tests (including computerized test) and interviews.
* Gave informed consent for participation in the study.

Exclusion Criteria:

* Dizziness disease with fluctuating symptoms such as in active Meniere's disease or Benign Paroxysmal Positional Vertigo
* CNS disease or injuries
* Dizziness caused as a result of previous whiplash
* Any active or non-controlled disease that might cause dizziness (e.g. non-controlled diabetes, hypertension, anemia, respiratory, cardiovascular or endocrinological disorder etc.)
* Pregnant women
* Participation currently in another clinical study or enrolled in another clinical study within 30 days prior to this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | After 4 weeks of treatment
  The change from baseline in dizziness symptoms as measured by Dizziness Handicap Inventory (DHI)
  The change from baseline in balance as measured by the Activities-specific and Balance Confidence (ABC) Scale.
  Safety:AE incidence Physical, neuro-otologic and neurological examination Static/dynamic/positioning examination

SECONDARY OUTCOMES:
Vertigo Symptom Scale-Short Form | After 4 weeks of treatment
  Vertigo Symptom Scale-Short Form
Visual Vertigo Analog Scale (VVAS) | After 4 weeks of treatment
  Visual Vertigo Analog Scale (VVAS)
The Activities-specific Balance Confidence (ABC) Scale | After 4 weeks of treatment
  The Activities-specific Balance Confidence (ABC) Scale
Clinical Global Impressions-Improvement (CGI-I) scale | After 4 weeks of treatment
  Clinical Global Impressions-Improvement (CGI-I) scale
Berg Balance Scale (BBS) | After 4 weeks of treatment
  Berg Balance Scale (BBS)
Beck Anxiety Inventory (BAI) | After 4 weeks of treatment
  Beck Anxiety Inventory (BAI)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gordon, Prof, Principal Investigator — Meir Medical Center
Locations (1):
- Dept Neurology, Meir Medical Center, Kfar Saba, Israel